CLINICAL TRIAL: NCT05779332
Title: Prevalence, Etiology and Effects on Oral Health and Life Quality of Molar Incisor Hypomineralization: A Comprehensive Study
Brief Title: Prevalence, Etiology and Effects on Oral Health and Life Quality of Molar Incisor Hypomineralization
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Aydınoglu, associate professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 140
Record Dates: First submitted 2023-01-19; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Molar Incisor Hypomineralization; Oral Health; Child, Only; Pediatric ALL; Dental Caries; Dental Plaque; Dental Diseases
Keywords: Molar Incisor Hypomineralization; oral health; MIH; Oral health related lif quality; Child Perceptions Questionnaire; OHRQoL; CPQ
MeSH Terms: conditions — Molar Hypomineralization; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dental Caries; Dental Plaque; Stomatognathic Diseases | interventions — Diagnosis, Oral

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey application — Children's OHRQoL was measured by the Child Perceptions Questionnaire (CPQ8-10). Oral examination of children were conducted for presence and severity of MIH, dental caries experience and oral hygiene status.
  Other Names: oral examination

SUMMARY:
Molar incisor hypomineralization (MIH) can lead to many clinical conditions and affect oral health-related quality of life (OHRQoL).

DETAILED DESCRIPTION:
Molar incisor hypomineralization (MIH) can lead to many clinical conditions and affect oral health-related quality of life (OHRQoL). The aim of this study was to determine the prevalence, etiology and impacts of MIH on oral health status and OHRQoL.

Six hundred and fifty-five parents and their children aged 9 years were included in the study. After parents completed the questionnaire about the etiology of MIH, children's OHRQoL was measured by the Child Perceptions Questionnaire (CPQ8-10). Children were evaluated for presence and severity of MIH, dental caries experience and oral hygiene status. Qualitative data were analyzed with the Pearson chi-square and Fisher's exact tests. For the quantitative data, if the normal distribution was not satisfied, Kruskal Wallis/Mann-Whitney U tests were used. Also, Binominal logistic regression analysis was performed and p<0.05 was statistical significant.

.

ELIGIBILITY:
Inclusion Criteria:

* Being 9-year-old,
* Mentally and physically capable of completing the questionnaire,
* Presence of fully erupted 4 permanent molars and 8 permanent incisors.

Exclusion Criteria:

* Children were receiving orthodontic treatment during the examination,
* Children had enamel hypoplasia or developmental defects,
* Children had amelogenesis imperfecta or dental fluorosis.

Ages: 9 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 9-year-old children who were enrolled in the primary schools in the city of Rize, Turkey.
Sampling Method: Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and etiology of MIH. | up to four months
  A questionnaire was applied to the parents about the etiological factors and the prevalence of MIH was determined by oral examination.
To evaluate the impacts of MIH on oral health status. | up to six months
  Oral health was evaluated by recording dmft (decayed, missing and filled teeth) and plaque index values.
To evaluate the impacts of MIH on OHRQoL. | up to six months
  The impact of MIH on quality of life (OHRQoL) was measured with the Child Perception Questionnaire (CPQ8-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Sema Aydinoğlu, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No